CLINICAL TRIAL: NCT04493073
Title: Comparison of Conjunctival Vascularity Changes Using Optical Coherence Tomography Angiography After Trabeculectomy With Mitomycin and Ologen Implants
Brief Title: Conjunctival Vascularity Changes Usnig OCTA After Trabeculectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asmaa Ahmed Ali Youssif (Other)
Responsible Party: Sponsor-Investigator, Asmaa Ahmed Ali Youssif, doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OCTA after Trabeculectomy
Record Dates: First submitted 2020-07-24; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: OCTA
MeSH Terms: interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trabectulectomy with mitomycin (Active Comparator): Mitomycin-C Kyowa® (Biochem Pharmaceutical Industries, India) 10 mg vial 2 mg/ml concentration
  Interventions: Procedure: Trabectulectomy; Drug: Mitomycin; Device: Mitomycin-C Kyowa®
- Trabectulectomy with Ologen implants (Active Comparator): Ologen Collagen Implant (Aeon Astron Europe, Netherlands) - three-dimensional collagen- GAG implant >90% lyophilized porcine atelocollagen and <10% lyophilized porcine GAG 12 mm in diameter with 1 mm of thickness and 6 mm in diameter with 2 mm of thickness
  Interventions: Procedure: Trabectulectomy; Device: Ologen Collagen Implant

INTERVENTIONS:
Procedure: Trabectulectomy — decrease IOP
Drug: Mitomycin — Decrease bleb failure
  Other Names: ologen implants
  Arms: Trabectulectomy with mitomycin
Device: Ologen Collagen Implant — Ologen Collagen Implant (Aeon Astron Europe, Netherlands)
  Arms: Trabectulectomy with Ologen implants
Device: Mitomycin-C Kyowa® — Mitomycin-C Kyowa® (Biochem Pharmaceutical Industries, India)
  Arms: Trabectulectomy with mitomycin

SUMMARY:
* Reduce the trauma and the time taken for patient rehabilitation.
* The prevailing trend is to perform a mitomycin- C (MMC)-augmented trabeculectomy and trabeculectomy with ologen implants in a trial to decrease bleb failure as a common post- trabeculectomy complication.
* Is to develop a measurement protocol by OCT-A imaging and characterization of the bleb vascularity changes in glaucoma patients before and after surgery.

DETAILED DESCRIPTION:
The main purpose of this project is to compare bleb vascularity changes using optical coherence tomography (OCT-A) between mitomycin- C (MMC)-augmented trabeculectomy and develop trabeculectomy with ologen implants to determine whether bleb vascularity measurements during preoperative and early postoperative periode could act as surrogate parameters to predict surgical outcomes.

Glaucoma often existent in the elderly population. Measuremets of bleb vascularity beginning to become an essential part of the glaucoma specialist's clinical and operative took. As investigators continue to collect data both clinically and in the laboratory, these various imaging modalities will shepherd surgeons into a more precise and predicable era of glaucoma surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years of age with primary or secondary open-angle glaucoma.
* Primary OAG (POAG) diagnosed on the basis of IOP measurements more than 21 mmHg, open angle on gonioscopy (Grade 3 or 4 on Schaffer grading system for angle width), glaucomatous visual field defects consistent with glaucomatous optic disc changes.
* PNAG was diagnosed by the presence of narrow or occludable angle on gonioscopy (Grade 2, or 1 on Schaffer grading system for angle width in at least 180° of the total circumference of the angle in primary position without indentation), glaucomatous optic disc changes, visual field defects and IOP more than 21 mmHg

Exclusion Criteria:

* pregnant or lactating female.
* previous intraocular surgery
* one-eyed patients.
* previous ocular trauma.
* uveitis-induced glaucoma, neovascular glaucoma, aphakic/pseudophakic glaucoma
* systemic connective tissue disease and missing more than 3 follow-up visits.
* Trabeculectomy augmented by either MMC or Ologen implant was indicated to study subjects if they had uncontrolled IOP under maximum antiglaucoma medications (3 antiglaucoma drugs) or due to poor socioeconomic status.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
conjunctival vascularity changes | 1 year
  conjunctival vascularity changes using OCTA

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Saad, Study Director — Assiut University

REFERENCES:
- [Background] He M, Wang W, Zhang X, Huang W. Ologen implant versus mitomycin C for trabeculectomy: a systematic review and meta-analysis. PLoS One. 2014 Jan 20;9(1):e85782. doi: 10.1371/journal.pone.0085782. eCollection 2014. PMID 24465704